CLINICAL TRIAL: NCT02116634
Title: Phase 1, 2 Study of Mesenchymal Stem Cells Injection in ALS (Amyotrophic Lateral Sclerosis) Patients
Brief Title: Mesenchymal Stem Cell Injection in Amyotrophic Lateral Sclerosis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Because economic problems
Sponsor: Alzahra Hospital, Iran (Other)
Responsible Party: Principal Investigator, rokhsareh meamar, Principal Investigator, Alzahra Hospital, Iran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rokhsareh; stem cell injection in ALS (Other: iran national science foundation)
Record Dates: First submitted 2014-04-06; First posted 2014-04-17 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mesenchymal stem cell (Experimental): intra spinal injection of 1 ×10(8) mesenchymal stem cells +10cc normal saline
  Interventions: Biological: mesenchymal stem cell

INTERVENTIONS:
Biological: mesenchymal stem cell — intra spinal injection of 1 ×10(8) mesenchymal stem cells +10cc normal saline

SUMMARY:
Whether the mesenchymal injection on ALS patients is effective or not?

DETAILED DESCRIPTION:
After and before transplantation, all of the patients will visit by experience neurologist and evaluate with EMG (electromyography) and spirometry procedure and clinical progression of disease.

ELIGIBILITY:
Inclusion Criteria:

1. sporadic ALS according to escorial criteria
2. onset of disease with spinal cord involvement, Less than 3 years of disease onset with disease progression at 6 past months
3. mild to moderate spinal and bulbar disability,at least having score3 in swallowing, 2 in chewing and waking in ALS-FRS and FVC(functional vital capacity) equal or more than 50% of prediction amount
4. normal polysomnography
5. Signed consent form

Exclusion Criteria:

1. pregnancy or lactation,
2. vascular disease,diabetes, systemic disease as cancer, autoimmune , liver or hematologic disease
3. Hospitalization due to serious illness in the last two months
4. survival time less than two years
5. Hypersensitivity to any component used in the cell culture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Effect of Intrathecal injection of autologous mesenchymal stem cells in improving the symptoms of ALS | every 6 months up 2 years after transplantation

SECONDARY OUTCOMES:
ALS-FRS(functional rating scale) score and EMG scale | before transplatation and at 6 months, 12months, 18 months and 24 months after transplantation
FVC (forced vital capacity)and DWSE±QoL score | before transplantation and every 6 months up 2 years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: keivan basiri, MD, Principal Investigator — Isfahan neurosciences research center
Locations (1):
- Neurosciences Research Center, Isfahan, Iran